CLINICAL TRIAL: NCT05108168
Title: Analysis of Clinical featuRes and Echocardiographic Characteristics for Diagnosis of Infiltrative cardiomyopaThy (ACREDIT): Retrospective Multi-center Observational Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2020-1278
Record Dates: First submitted 2021-10-24; First posted 2021-11-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Infiltrative Cardiomyopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- infiltrative cardiomyopathy: infiltrative cardiomyopathy

SUMMARY:
This study sought to develop an algorithm by collecting echocardiographic image information and related clinical information capable of quantitatively evaluating changes of the myocardium through machine learning. Moreover, the researchers investigate the usefulness of an algorithm for early diagnosis and differential diagnosis of infiltrative cardiomyopathy.

DETAILED DESCRIPTION:
1. Study Design: Multicenter Retrospective Observational Study
2. Study method: If the above selection criteria are met, the index visit echocardiographic images which were performed immediately before or closest to the time of hospitalization for final diagnosis, echocardiographic images of the pre-visit and post-visit from the final diagnosis, and clinical information will be obtained. Chest X-ray, electrocardiogram, and echocardiography images are extracted in raw DICOM format and then analyzed in the core lab (Severance hospital). The characteristics of patients with infiltrative cardiomyopathy are identified through the collection of relevant clinical information, and a method for non-invasive early diagnosis and differential diagnosis of infiltrative cardiomyopathy is developed.
3. Quantative analysis of echocardiographic images using Radiomics

   * Radiomics is a method of extracting a large number of quantitative image features (300-500 features such as shape, entropy, volume, etc.) from non-invasive medical images (CT, MRI, etc.) and statistically analyzing the features. Its value has been demonstrated through the studies for prediction of breast cancer recurrence and lesion classification.
   * Using the open source platform PyRadiomics19, we extract the radiomic characteristics for brightness (Energy, Entropy, Mean, Median, etc.) and texture (Gray Level Co-occurrence Matrix Contrast, Difference Variance, Maximal Correlation Coefficient, etc.) from the set region of interest.
   * The differences between infiltrative cardiomyopathy and normal control are identified using clinical information and radiomics features extracted from echocardiography at the time of the diagnosis visit. The algorithms to distinguish the disease will be developed using machine learning methods such as support vector machine classifier.

ELIGIBILITY:
Inclusion/exclusion criteria

1. Selection criteria for screening (1) 18 years old or older (2) Patients with infiltrative cardiomyopathy (the diagnostic name for each of the following diseases) or systemic disease (such as amyloidosis, multiple myeloma, sarcoidosis) (3) Search Period: January 1, 2010-December 31, 2020
2. Criteria for enrolling patients

   * Patients who are satisfied with at least one of each definition are selected.

     * Cardiac amyloidosis1,5,11,12 I. 'Definite': Positive myocardial biopsy (Congo-Red positive) II. 'Probable': One of the following imaging findings along with a positive biopsy of tissues other than myocardium A. Positive DPD / PYP scan Grade 2-3 cardiac uptake B. Echocardiography Symmetrical increase in LV and RV wall thickness Dilated LA and RA Granular appearance of myocardium Pericardial effusion Decreased or normal RQS complex voltage despite increased LV wall thickness C. Cardiac magnetic resonance imaging Diffuse subendocardial late Gd-enhancement Elevated native T1 and ECV value III. 'Possible': Two or more of the above imaging findings are satisfied without biopsy findings, and it is suitable for the diagnosis according to all clinical findings

       ② Cardiac sarcoidosis13,14,15,16 I. 'Definite': If all of the following are satisfied A. Noncaseating, multinucleated giant cell granuloma surrounded by bands of dense collagen fibers in endomyocardial biopsy B. Compatible clinical presentation C. Exclusion of other causes of granulomatous inflammation II. 'Probable': Two or more of the following findings along with a positive biopsy of tissues other than myocardium A. Electrocardiogram High-grade atrioventricular block (including complete atrioventricular block) or fatal ventricular arrhythmia (e.g., sustained ventricular tachycardia and ventricular fibrillation) B. Echocardiography Variable focal LV wall thinning (frequently at the basal septum, lateral wall) Focal wall motion abnormalities do not match coronary artery territory C. Cardiac magnetic resonance imaging Patch, basal and lateral LV wall late Gd-enhancement D. Positron Emission Tomography - Computed Tomography Focal increased FDG-uptake IV. 'Possible': Two or more of the above imaging findings are satisfied without biopsy findings, and it is suitable for the diagnosis according to all clinical findings
       * Hemochromatosis 17 I. 'Definite': Positive myocardial biopsy Iron deposits within the myocyte II. 'Probable': Non-myocardial tissue biopsy positive or iron overload clinical evidence (such as hereditary hemochromatosis, transfusion-dependent anemia) and the following imaging findings A. Echocardiography Dilated LV with global systolic dysfunction B. Cardiac magnetic resonance imaging Low T2* value of myocardium

   Etc

   ① Fabry disease18,19 I. 'Definite': Positive myocardial biopsy Enlarged myocytes with clusters of concentric glycolipid (myelinoid bodies) within lysosomes II. 'Probable': A-galactosidase A screening test and X-linked genetic test positive, along with the following echocardiographic findings A. Echocardiography Symmetrical increase in LV and RV wall thickness

   ② Danon disease20 I. 'Definite': Positive for genetic testing or biopsy of myocardial tissue, along with the following echocardiographic findings Symmetrical increase in LV and/or RV wall thickness Decreased LV systolic function

   ③ Cardiac oxalosis1 I. 'Definite': Positive myocardial biopsy II. 'Probable': The following echocardiographic findings along with a history of massive transfusion or positive biopsy of tissues other than myocardium Symmetrical increase in LV and RV wall thickness Patchy, echodense speckled reflection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is important to obtain as large image data as possible to develop an algorithm capable of diagnosing various infiltrative myocardial diseases.
  Infiltrative cardiomyopathy is a rare disease, and it was reported that the prevalence of cardiac amyloidosis in Korea was 1.91 per 100,000 in 2015.2 In the case of other diseases, there has been no report of the prevalence in Korea, but reports from an overseas report that cardiac sarcoidosis is 2.2 per 100,000, 8 and Fabry disease is 0.9 to 2.5 per 100,000. 9,10 Securing enough data that can be learned to improve machine learning accuracy is not easy because of the scarcity of invasive cardiomyopathy. Furthermore, it is difficult to confirm the disease. Therefore, it is necessary to review and obtain clinical information and echocardiographic image data of as many confirmed patients as possible. This study is a retrospective observational study, and the expected number of target subjects is about 500.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-01-04 (Actual); Primary Completion 2021-12-16 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | until June 30, 2022
  Sensitivity (True Positive Rate) refers to the proportion of those who have the infiltrative cardiomyopathy that received a positive result on the diagnostic algorythm by machine learning.
Specificity | until June 30, 2022
  Specificity refers to the proportion of those who do not have the infiltrative cardiomyopathy that received a negative result on the test.
Area under the curve of the receiver operation characteristics | until June 30, 2022

CONTACTS AND LOCATIONS:
Overall Officials: Hyuk-jae Chang, Principal Investigator — Yonsei University Health System, Severance Hospital, Division of Cardiology
Locations (1):
- Yonsei University Health System, Severance Hospital, Division of Cardiology, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seward JB, Casaclang-Verzosa G. Infiltrative cardiovascular diseases: cardiomyopathies that look alike. J Am Coll Cardiol. 2010 Apr 27;55(17):1769-79. doi: 10.1016/j.jacc.2009.12.040. PMID 20413025
- [Background] van Griethuysen JJM, Fedorov A, Parmar C, Hosny A, Aucoin N, Narayan V, Beets-Tan RGH, Fillion-Robin JC, Pieper S, Aerts HJWL. Computational Radiomics System to Decode the Radiographic Phenotype. Cancer Res. 2017 Nov 1;77(21):e104-e107. doi: 10.1158/0008-5472.CAN-17-0339. PMID 29092951